CLINICAL TRIAL: NCT01787669
Title: A Multicentre Clinical Trial of Switching Between Intravitreal Bevacizumab (Avastin®) and Intravitreal Dexamethasone (Ozurdex™) for Persistent Diabetic Macular Oedema (SwitchDMO)
Brief Title: Trial of Switching Between Intravitreal Bevacizumab (Avastin®)& Intravitreal Dexamethasone (Ozurdex™) for Persistent Diabetic Macular Oedema
Acronym: SwitchDMO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SwitchDMO
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Diabetes; Diabetic Macular Oedema; Diabetic Macular Edema; Diabetic Retinopathy
Keywords: diabetic macular oedema; diabetic macular edema; diabetic retinopathy; dexamethasone; Ozurdex; Avastin; bevacizumab; DME; DMO
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy | interventions — Bevacizumab; Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Avastin (bevacizumab) (Active Comparator): Intravitreal Avastin loading doses followed by as prn for remainder of 6 months according to defined retreatment criteria
  Interventions: Drug: Avastin (Bevacizumab)
- Ozurdex (dexamethasone) (Active Comparator): single dose at baseline and repeat dose when required according to defined re-treatment criteria
  Interventions: Drug: Ozurdex (dexamethasone)

INTERVENTIONS:
Drug: Avastin (Bevacizumab) — Avastin (Bevacizumab) administered intravitreally
  Arms: Avastin (bevacizumab)
Drug: Ozurdex (dexamethasone) — Ozurdex (dexamethasone) given intravitreally
  Arms: Ozurdex (dexamethasone)

SUMMARY:
The specific aim of the study is to test the following hypothesis:

That switching between treatments from bevacizumab to Ozurdex or vice versa in eyes with diabetic macular oedema with no or incomplete response from one therapy is beneficial.

DETAILED DESCRIPTION:
A Multicentre Clinical Trial of Switching Between Intravitreal Bevacizumab (Avastin®) and Intravitreal Dexamethasone (Ozurdex™) for Persistent Diabetic Macular Oedema (SwitchDMO)

ELIGIBILITY:
Inclusion Criteria:

Eyes Previously Treated with bevacizumab:

1. Diabetic macular oedema affecting the fovea that has persisted despite ongoing, monthly intravitreal injections of bevacizumab over at least 6 months, the last being 2 to 3 months prior to the screening visit.
2. There must be an historical OCT available from 1-4 weeks after the last bevacizumab injection with retinal thickness > 300 microns in the central 1mm subfield on Spectral domain OCT to show the lack of complete response to bevacizumab.
3. At screening, the bevacizumab treated eye must have DMO with retinal thickness > 300 microns in the central 1mm subfield on Spectral domain OCT

   Eyes Previously Treated with dexamethasone:
4. Diabetic macular oedema affecting the fovea that has persisted despite two dexamethasone implants 5 or fewer months apart, the last being 5-8 months prior to the screening visit.
5. There must be an historical OCT available from 8-14 weeks after the last dexamethasone implant with retinal thickness > 300 microns in the central 1mm subfield on Spectral domain OCT to show the lack of complete response to the dexamethasone implant.
6. At screening, the dexamethasone treated eye must have DMO with retinal thickness > 300 microns in central 1mm subfield on Spectral domain OCT
7. Age >= 18 years
8. Diagnosis of diabetes mellitus
9. Best corrected visual acuity of 20-78 letters (approx 6/120 -6/7.5)
10. Previous macular laser treatment, or the investigator believes laser treatment is unlikely to be helpful
11. Intraocular pressure <22mmHg
12. Women of childbearing potential must have a negative urine pregnancy test at the screening visit and prior to treatment. A woman is considered of childbearing potential unless she is postmenopausal and without menses for 12 months or is surgically sterilised
13. Written informed consent has been obtained.

Exclusion Criteria:

* Treatment with intravitreal triamcinolone acetonide (IVTA) within the last 6 months or peribulbar TA within the last 3 months, or anti vascular endothelial growth factor (VEGF) drugs: ranibizumab and aflibercept, within the last 2 months.
* Cataract surgery within the last 3 months
* Retinal laser treatment within the last 3 months
* For eyes to be switched to Dexamethasone: Patient considered, at the judgement of the investigator, to be at-risk for syphilis, tuberculosis or other potentially infective chorioretinopathies. Patients considered at-risk may be assessed at the investigators discretion to reasonably exclude these conditions. Should these conditions be excluded, the patient may be considered for enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-06; Primary Completion 2017-01 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Proportion of eyes that have central macular thickness <300 microns 6 months after switching | 6 months

SECONDARY OUTCOMES:
Mean change in central macular thickness (CMT) as measured by OCT. | 6 months
  Mean change in central macular thickness (CMT) as measured by OCT.

OTHER OUTCOMES:
Mean change in BCVA (best corrected visual acuity) | 6 months
  Proportion of eyes with a gain of 15 LogMAR letters or more
  * Proportion of eyes with a loss of less than 15 LogMAR letters
  * Proportion of eyes with gain of 5 LogMAR letters or more
  * Proportion of eyes with gain of 10 LogMAR letters or more

CONTACTS AND LOCATIONS:
Overall Officials: Samantha FRASER-BELL, Principal Investigator — SAVE SIGHT INSTITUTE, UNIVERSITY OF SYDNEY, SYDNEY EYE HOSPITAL
Locations (3):
- Australia (3):
  - Sydney Eye Hospital, Sydney, New South Wales
  - Centre for Eye Research Australia (Royal Victorian Eye & Ear Hospital), Melbourne, Victoria
  - Lions Eye Institute, Perth, Western Australia